CLINICAL TRIAL: NCT06560567
Title: Investigation of the Attitudes and Barriers of Prosthetics and Orthotics Professionals in Turkey Towards 3D Printers and Technology
Brief Title: Attitudes and Barriers of Prosthetics and Orthotics Professionals in Turkey Towards 3D Printers and Technology
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ayse Yazgan, Lecturer, Medipol University
Other Study IDs: MedipolU-OP-AY-02
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Technology
Keywords: Three-Dimensional Printing; Anxiety; Orthosis; Limb prosthesis
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prosthetics and Orthotics Professionals: A total of 131 participants, 29 female and 102 male, aged at least 18 and at most 65 years old, completed the survey. The inclusion criteria for the participants were determined as working in an Orthosis and Prosthesis Application Center and being 18 years of age or older.

SUMMARY:
This study aim is the attitudes and barriers of prosthetics and orthotics professionals towards 3D printers and technology will be determined.

DETAILED DESCRIPTION:
It is known that there are generally concerns about high capital costs and return on investment in the use of 3D printer technology in Turkey.

It is known that there is no study in Turkey to investigate the attitudes and barriers of prosthetics and orthotics professionals towards 3D printers and technology. Therefore, the attitudes and barriers of prosthetics and orthotics professionals towards 3D printers and technology will be questioned in the study. It was aimed to reveal the perspectives and concerns about 3D printers and technology and to emphasize the importance of increasing the number of education and competent personnel regarding the dissemination of technological applications in practice.

In the study investigating the attitudes and barriers of prosthetics and orthosis professionals towards 3D printers and technology in Turkey, a total of 131 participants, 29 female and 102 male, aged at least 18 and at most 65 years old, were included.

The participants first filled out the Demographic Information Form. This form includes demographic information such as the participant's age, gender, education level, profession, duration of professional experience, geographical region where they work, the number of in-service trainings they receive in the field of orthosis and prosthesis, weekly working hours and the number of daily patients they communicate with.

At the end of the demographic information, the participants were asked to state open-endedly what they had concerns about technology that they could not define.

In addition, questions created according to the Technology Acceptance Model (TAM) and the Affinity for Technology Interaction (ATI) were also answered by the participants.

When the participants were asked whether they had concerns about 3D printers and technology that they could not define, it was determined that they mostly answered no. When the participants who had concerns were asked open-endedly about their concerns, the answers given were mostly about the lack of information or competent personnel for use when the answers were collected under common headings. It was observed that the technology acceptance model and proximity to technology had an effect on the time spent in the profession and the total score of ATI.

ELIGIBILITY:
Inclusion Criteria:

* As working in an Orthosis and Prosthesis Application Center
* Being 18 years of age or older.

Exclusion Criteria:

* Insufficient cognitive level to answer the survey

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 131 participants, 29 female and 102 male, aged at least 18 and at most 65 years old, completed the survey. The inclusion criteria for the participants were determined as working in an Orthosis and Prosthesis Application Center and being 18 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Technology Acceptance Model (TAM) | immediately after screening
  While creating the TAM survey, a total of 23 questions were asked to measure the perceived of usefulness, perceived ease of use, attitude variable, intention variable and the behavior variable towards 3D Printing and Technology.
  Questions were also asked to determine demographic characteristics. Demographic information questions are; participant's age, gender, education level, job, work experience (years), job geographic region, number of in-service trainings in orthotics and prosthetics, weekly working hours and number of patients contacted daily. At the end of the demographic information, participants were asked to clearly state their concerns about technology that they could not define.
  While the questions regarding demographic targets in the survey were categorical, the questions measuring perceptions regarding the use of 3D printing and technology included 5-point Likert type answers. (1: Strongly disagree, 2: Disagree, 3: Neutral, 4: Agree, 5: Strongly agree)
Affinity for Technology Interaction (ATI) | immediately after screening
  ATI evaluates the affinity to technology by focusing on user-system interaction. The scale takes into account cognitive needs to base affinity to technology on basic psychological structures and the questions are formulated accordingly. The title of the scale includes the statement that questions will be asked about interaction with technical systems. In our study, 3D Printer technology was stated to the participants as a technical system. The scale consists of 9 questions and the answers are in the form of a 6-point Likert scale: '1=Totally disagree, 2=Mostly disagree, 3=Partially disagree, 4=Partially agree, 5=Mostly agree, 6=Totally agree'. Finally, an average score was calculated over the 9 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Yazgan, Principal Investigator — https://www.medipol.edu.tr/
Locations (1):
- Ayşe Yazgan, Bakırköy, Istanbul, Turkey (Türkiye)